CLINICAL TRIAL: NCT05622825
Title: Evaluation of the Safety and Efficacy of Combination of Cryoablation and Dendric Cell/Cytokine-induced Killers Cells Treatment for Advanced Liver Cancers
Brief Title: Valuation of the Safety and Efficacy of Combination of Cryoablation and Dendric Cell/Cytokine-induced Killers Cells Treatment for Advanced Liver Cancers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202112056DIPC
Record Dates: First submitted 2022-10-13; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Advanced Liver Cancers
Keywords: DC-CIK; Cryoablation; Advanced Liver Cancers

STUDY DESIGN:
Intervention Model Description: Patients must receive 2 DC/AT hepatic artery infusion and be treated with cryoablation technique.
  Phase Ⅰ The first 3 subjects were enrolled by Sequential enrollment. The next subject can be enrolled only after the first subject has completed the return transfusion and the safety assessment (V7). After the sixth subject completes the safety assessment (V7), the next nine subjects can be enrolled in phase IIA of the trial to evaluate the efficacy of the trial. If less than two of the first six subjects have a Common Terminology Criteria for Adverse Events (CTCAE) v5.0 level 3 or higher adverse event related to the test drug Phase Ⅱ Phase IIA to evaluate the efficacy and implementation. However, if two of the first six subjects have a Grade 3 or higher trial drug-related adverse event or one or more deaths, the trial will be terminated immediately and all cell product process-related factors in this trial will be fully investigated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cryoablation combined DC-CIK (Experimental): To explore the therapeutic effect and safety of cryoablation combined with autologous DC-CIK (through hepatic artery infusion, HIA) for patients with advanced liver cancers
  Interventions: Biological: DC-CIK

INTERVENTIONS:
Biological: DC-CIK — To explore the therapeutic effect and safety of cryoablation combined with autologous DC-CIK (through hepatic artery infusion, HIA) for patients with advanced liver cancers

SUMMARY:
The treatment of liver cancer needs integrated medical strategies, including surgery, chemotherapy, target therapy, radiotherapy, and immunotherapy. According to the patient's condition to develop a personalized and best treatment plan. Cryoablation can produce osmotic shock through repeated freeze-thaw to cause tumor cell necrosis, and release tumor antigens to activate anti-tumor immune responses. Immune cell therapy is an emerging field across cancer types in current cancer treatment. This study desired to combine cryotherapy and cellular immunotherapy to achieve the effect of tumor control. In recent years, cancer treatment studies have showed that cryoablation combined with immune cell therapy can play a good auxiliary effect and improve the cancer treatment efficacy significantly.

This trial study is a single center, single-arm, non-blind open-label human clinical trial. To explore the therapeutic effect and safety of cryoablation combined with autologous DC-CIK (through hepatic artery infusion, HAI) for patients with advanced liver cancers. The DC-CIK biologics are provided by BOHUI Biotech company. Their core technology (including clinical treatment and cell culture techniques) was transferred from Dr. Hasumi who is a Japanese clinician and this technical founder.

DETAILED DESCRIPTION:
The World Health Organization's International Agency for Research on Cancer (IARC) has released the latest global cancer burden data for 2020, which shows that 19.3 million new cancer cases happened and nearly 10 million deaths occurred in 2020. Currently, one in five people of the world will have cancer in their lifetime, and one in eight men and one in 11 women will die of cancer. According Taiwan Cancer registry introduction from Ministry of Health and Welfare in 2017, the number of new cancer cases was 111,684, 5,852 more people than in 2015. Liver cancer, in particular, ranks fourth in the cancer rankings. The main causes of liver cancer are hepatitis B, hepatitis C, or cirrhosis of the liver caused by alcohol. Other causes include Aspergillus flavus toxin, non-alcoholic fatty liver disease and liver aspirates etc.

Immune cell therapy is an emerging field in the treatment of advanced liver cancer. Many types of immune effector cells such as lymphokine-activated killer (LAK) cells, dendritic cells (DC), tumor infiltrating lymphocyte (TIL) cells, cytokine-induced killer (CIK) cells, and lymphocyte-activated lymphocyte (LAK) cells are used to treat advanced liver cancer. CIK cells have been developed for immunotherapy applications. CIK cells such as CD3+CD56+ cells, CD3+CD56- cells and CD3-CD56+ cells, have the ability to kill tumors directly by demonstrating the non-restrictive cytolytic effect of MHC, similar to the function of general T cells. CIK cells bind to LFA-1 ligands on tumor cells through LFA-1, resulting in tumor cell killing, and then binding of the receptor to its ligand on NK cells initiates a downstream cell signaling pathway and further activates CIK cells for tumor cytotoxicity. Finally, CIK cells activate the signaling pathway via Fas-FasL and induce apoptosis in cancer cells. DCs are differentiated from hematopoietic stem cells in the bone marrow, often in the form of monocytes, which differentiate into mature dendritic cells in response to cytokine stimulation. After tumor-associated antigen (TAA) phagocytosis, antigens are treated by two pathways, the cytosolic pathway and vacuolar pathway, by which they are processed into peptides and loaded onto the major histocompatibility complex class I(MHC I). Then the TAA-MHC I complex is delivered to the DC surface. When DC-presenting TAAs migrate and reach the lymph nodes, they are able of priming T cells and prompting anti-tumor immunity. Dendritic cells are efficient activators of naïve T cells and are potent APCs. They play a central role in immune-mediated cancer elimination through antigen presentation and T-cell priming. More recently, they have been combined to form DC-CIK cell therapy, which is a combination immunotherapy where DC and CIK cells are cultured together. In terms of therapeutic mechanism, dendritic cells are specialized antigen-presenting cells, and mature dendritic cells can present tumor antigens via the MHC-I pathway to effectively counteract the immune escape mechanism of tumor cells. The specific tumor-killing effect of CIK is further enhanced. Many studies have shown that treating cancer patients with DC-CIK cells significantly prolong the survival time and enhance the immune function of the patient.

Recent trends in cancer treatment have confirmed that when cryoablation of tumors is combined with immune cell therapy, it can have a good complementary effect and significantly improve the efficacy of cancer treatment. It is believed that cryotherapy causes necrosis of tumor cells through the physical changes of osmotic shock produced by repeated freezing and thawing, which in turn releases tumor antigens and activates anti-tumor immune responses. A retrospective study conducted in 2013 in patients with stage IV lung cancer investigated the efficacy of cryoablation combined with immune cell DC-CIK and showed that cryoablation with DC-CIK significantly prolonged the overall survival (OS) of patients. The results of the 2017 clinical trial showed that cryoablation with NK cell therapy improved the clinical response rate and disease control rate (DCR) of patients with advanced lung cancer, with the proportion of patients with PR (63.3% vs. 43.3%, P<0.01) and disease control rate ( The results of the clinical trial in advanced hepatocellular carcinoma showed that among 61 patients admitted from 2015 to 2017, cryoablation with NK immunotherapy significantly prolonged the progression free survival (PFS) of patients (9.5%). (PFS) (9.1 months vs. 7.6 months, P=0.0107), response rate (60% vs. 46.1%, P<0.05) and disease control rate (85.7% vs. 69.2%, P<0.05).

The trial was designed as a single-arm, uncontrolled, open-label, non-random assignment design. The efficacy and safety of hepatic artery infusion with autologous DC-CIK immune cells before and after ablation of liver tumors using cryoablation technique in patients with advanced liver cancer was investigated. The DC-CIK immune cell therapy technology was developed in collaboration with Bohui Biotech, and the core cell technology was transferred from Dr. Hasumi autologous immune cell therapy in Japan. The program will track the changes in tumor size and tumor index before and after treatment, and conduct safety assessment to evaluate the safety and efficacy of this trial treatment.

During the clinical trial, peripheral blood will be collected from patients for exploratory index analysis to complement the clinical evaluation results. According to the results of the clinical study in 2013, patients with stage IV solid cancer who had failed standard treatment had increased CD8+CD56+ cell populations after autologous immune cell therapy by Dr. Hasumi in Japan and continued to be followed up until one year later. In 2019, a study also showed that disease control was lower in the group of patients with liver cancer with high free DNA concentrations treated with sorafenib than in the group with low free DNA concentrations. The whole-genome sequencing of cell-free DNA (cfDNA) to obtain copy number alteration (CNA) profiles can be used as predictors of sorafenib treatment outcome. Therefore, in this clinical trial, blood samples were taken from patients before and after treatment, and the distribution of immune cell populations and changes in cell-free DNA (cfDNA) in blood were analyzed separately by separating the buffy coat and plasma using a density gradient centrifuge, and using the Qubit 2.0 Fluorometer. The qubit dsDNA High Sensitivity assay kit (Life Technology, Carlsbad, CA, USA) was used to quantify the amount of free DNA and to detect the copy number of free DNA, and to analyze the free DNA to find out the biomarkers that can be used for treatment effect tracking.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 and 80 years old.
2. Patients with advanced stage hepatocellular carcinoma or advanced stage hepatic metastasis derived from extrahepatic primary carcinoma, who are judged as advanced stage by clinical criteria (The Eighth Edition AJCC Cancer Staging Manual) through pathology and imaging reports.
3. Patients who have been evaluated by a physician for benefits and risks and are no longer considered suitable for previous third-line therapies will be included in this trial.
4. There is at least one target lesion larger than 1.0 cm that can be measured by MRI or CT and is appropriately located for cryoablation by imaging.
5. Child-Pugh class (A or B).
6. Adequate bone marrow function (white blood cell count > 2x109/L, platelet count > 5x1010/L).
7. coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal
8. renal function: blood creatinine concentration (creatinine) < 1.5 mg/dL .
9. Karnofsky Performance Status (KPS) score70 -10.
10. maximum tumor diameter ≤ 5 cm
11. number of tumors ≤ 5
12. Survival period greater than 3 months as predicted by the physician.

Exclusion Criteria:

1. Tumor size >5 cm in diameter or tumor number >5.
2. not suitable for cytarabine or cryoablation as determined by the trial physician.
3. Blood screening for any of the following viral infections: human immunodeficiency virus, human T-lymphotropic virus, syphilis, hepatitis B virus, hepatitis C virus, cytomegalovirus IgM antibody positive, etc.
4. Previous treatment prior to screening: Chemotherapy or radiation therapy must be completed before 3 weeks of screening to avoid systemic immune responses interfering with the immune cell therapy. If participating in clinical trials of other biologic agents or immunotherapy, at least 4 weeks of screening is required.
5. Patient is acutely or chronically infected or in acute cytomegalovirus attack at the time of screening.
6. Patients with level 3 hypertension, or patients with severe coronary disease.
7. patients with autoimmune disease.
8. patients who are pregnant, breastfeeding, or unable to use effective contraception.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Image Assessment | 6 weeks after treatment
  Evaluation of the treatment outcome using computed tomography (CT or PET/CT) or magnetic resonance imaging (MRI) to facilitate comparison of pre- and post-treatment differences. Response Evaluation Criteria in Solid tumor (RECIST criteria) will be used to evaluate the treatment effect of target lesions after treatment. The RECIST criteria will calculate Disease Control Rate.

SECONDARY OUTCOMES:
Quality of life assessment. | 12 weeks after treatment
  Pre- and post-treatment Eastern Cooperative Oncology Group (ECOG) measures changes in values. The overall physical health and quality of life is scored on normal, no complaints(0) to dead(5)
Quality of life assessment. | 12 weeks after treatment
  Pre- and post-treatment Cancer Quality of Life Questionnaire (EORTC QLQ- C30 Chinese version 3) measures changes in values. The overall physical health and quality of life is scored on a 7-point scale from very poor (0) to very good (7)

REFERENCES:
- [Background] Yun YS, Hargrove ME, Ting CC. In vivo antitumor activity of anti-CD3-induced activated killer cells. Cancer Res. 1989 Sep 1;49(17):4770-4. PMID 2527087
- [Background] Schmidt-Wolf IG, Negrin RS, Kiem HP, Blume KG, Weissman IL. Use of a SCID mouse/human lymphoma model to evaluate cytokine-induced killer cells with potent antitumor cell activity. J Exp Med. 1991 Jul 1;174(1):139-49. doi: 10.1084/jem.174.1.139. PMID 1711560
- [Background] Schmidt-Wolf IG, Lefterova P, Mehta BA, Fernandez LP, Huhn D, Blume KG, Weissman IL, Negrin RS. Phenotypic characterization and identification of effector cells involved in tumor cell recognition of cytokine-induced killer cells. Exp Hematol. 1993 Dec;21(13):1673-9. PMID 7694868
- [Background] Pievani A, Borleri G, Pende D, Moretta L, Rambaldi A, Golay J, Introna M. Dual-functional capability of CD3+CD56+ CIK cells, a T-cell subset that acquires NK function and retains TCR-mediated specific cytotoxicity. Blood. 2011 Sep 22;118(12):3301-10. doi: 10.1182/blood-2011-02-336321. Epub 2011 Aug 5. PMID 21821703
- [Background] Cappuzzello E, Sommaggio R, Zanovello P, Rosato A. Cytokines for the induction of antitumor effectors: The paradigm of Cytokine-Induced Killer (CIK) cells. Cytokine Growth Factor Rev. 2017 Aug;36:99-105. doi: 10.1016/j.cytogfr.2017.06.003. Epub 2017 Jun 3. PMID 28629761
- [Background] Lu PH, Negrin RS. A novel population of expanded human CD3+CD56+ cells derived from T cells with potent in vivo antitumor activity in mice with severe combined immunodeficiency. J Immunol. 1994 Aug 15;153(4):1687-96. PMID 7519209
- [Background] Yakkala C, Chiang CL, Kandalaft L, Denys A, Duran R. Cryoablation and Immunotherapy: An Enthralling Synergy to Confront the Tumors. Front Immunol. 2019 Sep 24;10:2283. doi: 10.3389/fimmu.2019.02283. eCollection 2019. PMID 31608067
- [Background] Yuanying Y, Lizhi N, Feng M, Xiaohua W, Jianying Z, Fei Y, Feng J, Lihua H, Jibing C, Jialiang L, Kecheng X. Therapeutic outcomes of combining cryotherapy, chemotherapy and DC-CIK immunotherapy in the treatment of metastatic non-small cell lung cancer. Cryobiology. 2013 Oct;67(2):235-40. doi: 10.1016/j.cryobiol.2013.08.001. Epub 2013 Aug 13. PMID 23948179
- [Background] Liu Y, Liu H, Liu H, He P, Li J, Liu X, Chen L, Wang M, Xi J, Wang H, Zhang H, Zhu Y, Zhu W, Ning J, Guo C, Sun C, Zhang M. Dendritic cell-activated cytokine-induced killer cell-mediated immunotherapy is safe and effective for cancer patients >65 years old. Oncol Lett. 2016 Dec;12(6):5205-5210. doi: 10.3892/ol.2016.5337. Epub 2016 Nov 2. PMID 28105230
- [Background] Lin M, Liang SZ, Wang XH, Liang YQ, Zhang MJ, Niu LZ, Chen JB, Li HB, Xu KC. Clinical efficacy of percutaneous cryoablation combined with allogenic NK cell immunotherapy for advanced non-small cell lung cancer. Immunol Res. 2017 Aug;65(4):880-887. doi: 10.1007/s12026-017-8927-x. PMID 28508945
- [Background] Hasumi K, Aoki Y, Wantanabe R, Mann DL. Clinical response of advanced cancer patients to cellular immunotherapy and intensity-modulated radiation therapy. Oncoimmunology. 2013 Oct 1;2(10):e26381. doi: 10.4161/onci.26381. Epub 2013 Oct 17. PMID 24349874
- [Background] Oh CR, Kong SY, Im HS, Kim HJ, Kim MK, Yoon KA, Cho EH, Jang JH, Lee J, Kang J, Park SR, Ryoo BY. Genome-wide copy number alteration and VEGFA amplification of circulating cell-free DNA as a biomarker in advanced hepatocellular carcinoma patients treated with Sorafenib. BMC Cancer. 2019 Apr 1;19(1):292. doi: 10.1186/s12885-019-5483-x. PMID 30935424